CLINICAL TRIAL: NCT03680118
Title: Vertical Ridge Augmentation Using Autogenous Onlay Ring Blocks Combined With Guided Bone Regeneration Using Collagen Membrane Versus Autogenous Bone Graft Only Using Titanium Mesh in Atrophic Posterior Mandibles.
Brief Title: Vertical Ridge Augmentation With Autogenous Onlay Blocks Combined With Guided Bone Regeneration Versus Autogenous Bone Graft With Titanium Mesh in Posterior Mandible
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Shawky Abd El-Moneim Shaheen, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cairouimplant masters
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Posterior Mandible With Deficient Ridge Height
MeSH Terms: interventions — Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- autogenous rings with GBR and autogenous graft with ti-mesh (Experimental): Augmentation with autogenous onlay ring blocks covered by guided bone regeneration (GBR) using collagen membrane and autogenous bone graft using titanium mesh (ti-mesh) only
  Interventions: Device: autogenous rings with GBR and autogenous graft with ti-mesh

INTERVENTIONS:
Device: autogenous rings with GBR and autogenous graft with ti-mesh — * Autogenous Onlay ring block harvested from either mandibular ramus or chin will be placed over the defected site and fixed using titanium screws (1.6mm diameter) and then GBR using autogenous particulate will be placed around and over the blocks and covered with a resorbable bilayer collagen membrane (Bio-Gide®, Geistlich, USA)
  * Autogenous bone graft will be placed on the defected site and covered by a titanium mesh which will be fixed by titanium screws.
  * Flap advancement will be acquired by releasing the mylohyoid muscle attachment from the lingual flap and periosteal releasing incision for the buccal flap to provide tension free closure.
  * The flap will then be copiously irrigated with saline in preparation for closure.
  * The flap will then be closed using horizontal mattress and interrupted 4/0 polypropylene sutures.

SUMMARY:
Atrophic ridge augmentation utilizing guided bone regeneration (GBR) has become a major treatment option to provide optimal bone support for osseointegrated dental implants. GBR was initially employed to treat simple defects, including dehiscence and fenestration defects. In addition, GBR has been utilized for horizontal and vertical ridge augmentations and has demonstrated reproducible outcomes, with high implant survival rates and low complication rates. The results of recent clinical and histologic studies of ridge augmentation with GBR indicated that autogenous bone graft may be a suitable material for staged localized ridge augmentation in both horizontal and vertical augmentations. The main advantages of autogenous grafts are their osteogenic, osteoinductive and osteoconductive capabilities. Because of these qualities, autogenous grafts are considered by many to be the gold standard for bone regeneration

DETAILED DESCRIPTION:
The GBR Procedure requires to place a barrier between the bone graft and the surrounding soft tissues. This blocks the fast-duplicating connective and epithelial cells from colonizing the regenerating site.

Collagen membranes have been successfully used as a barrier membrane in clinical practice.

They have the advantage of being resorbable and pose less post-operative complications. On the other hand, collagen membranes are not rigid, causing a difficulty in maintaining the vertical height of the particulate bone graft placed onto the ridge.

Alternatively, titanium meshes have been used with success in clinical practice and display both advantages and disadvantages. They provide tenting effect thanks to their rigidity and, being moldable, can be easily given the shape needed to cover the defect.

However they must be removed, not resorbable, require time-consuming shaping and pose complications as flap dehiscence.

Choice of the comparator:

Current studies have shown that using titanium mesh as a barrier to protect the bone graft during GBR can be considered successful in terms of vertical bone gain.

There might be variable in other findings which could be attributed to differences in the methodology, such as using other membranes over the titanium mesh (collagen or PTFE membranes).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with edentulous posterior mandible.
* Both sexes.
* No intraoral soft and hard tissue pathology.
* No systemic condition that contraindicate implant placement.
* Residual alveolar bone height more than 6 mm (7-9 mm) and less than 12 mm.

Exclusion Criteria:

* Presence of fenestrations or dehiscence of the residual ridge.
* Heavy smokers more than 20 cigarettes per day.
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-12-15 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
vertical bone gain | 6 month
  the amount of vertical bone gain will be measured using cone beam computed tomography